CLINICAL TRIAL: NCT05160844
Title: Association of SIRT1(rs7069102 ) Gene Polymorphism With Premature Myocardial Infarction in Young Egyptian Patients
Brief Title: SIRT1 Gene Polymorphism With Premature Myocardial Infarction in Young Egyptian Patients
Acronym: SIRT1
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amera Morad Foad, clinical professor, Sohag University
Other Study IDs: Soh-Med-21-11-33
Record Dates: First submitted 2021-12-06; First posted 2021-12-16 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Premature Myocardial Infarction in Young Egyptian Patients

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diseased: young Egyptian patients with premature myocardial infarction
- Control: healthy young Egyptians

SUMMARY:
This is an observertional study aimed at Study the association of SIRT1(rs7069102 ) Gene polymorphism with premature myocardial infarction in young Egyptian patients

ELIGIBILITY:
Inclusion Criteria:

* All patient with recent MI admitted to Sohag University Hospital , CCU under 40 years

Exclusion Criteria:

* patients above 40 year old.
* Patients with malignancies, major trauma or surgery in the previous six months, and acute or chronic infectious disease

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: young egyptian patients under 40 years of age presented with recent MI admitted to CCU at sohag university hospital.
Sampling Method: Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Endothelial nitric oxide synthase level | 6 months
  detect the serum level of Endothelial nitric oxide synthase by ELIZA in nanogram per millilitre (ng/ml)
SIRT1 Genotyping | 6 months
  whether homgenetic or heterogenetic

CONTACTS AND LOCATIONS:
Overall Officials: Amera Morad Foad hamdy, lecturer, Principal Investigator — Sohag faculty of medicine
Locations (1):
- Sohag uniersity hosoital, Sohag, Egypt